CLINICAL TRIAL: NCT01434771
Title: Simultaneous Hemodynamic and Ventilatory Monitoring Using Radio Frequency Impedance Interrogation (RFII), Thoracic Impedance Cardiography and Invasive Hemodynamic Monitoring Methods in Post Operative Cardiac Patients
Brief Title: Monitoring Blood Flow and Breathing Using a New Device (RFII) Compared to the Gold Standard Device in Post Operative Cardiac Patients
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor never funded study.
Sponsor: University of Florida (Other)
Collaborators: Noninvasive Medical Technologies, Inc. (Industry); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 20110031
Record Dates: First submitted 2011-09-13; First posted 2011-09-15 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Noninvasive Cardiac Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study will be to compare standard of care invasive methods to an FDA approved non-invasive device and a novel wireless non-invasive device, both manufactured by Non-Invasive Medical Technologies Inc., with the goal of correlating the data generated by the novel device to the measurements taken by the standard of care invasive monitors.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Weight - 36-136 Kilograms
* Height - 1.52 meters - 1.92 meters (5'- 6'4")
* Scheduled for open heart surgery during the study period

Exclusion Criteria:

* ECG lead adhesive allergy or sensitivity
* Pregnant Patients
* Prisoners
* Cognitively impaired
* Patients requiring mechanical cardiac support, or requirement for hemodialysis
* Patients not requiring pulmonary artery catheters for medical management.
* Patients with significant valvular disease will be enrolled if there is no significant post-repair valvular dysfunction as determined by intraoperative transesophageal echocardiography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for open heart surgery
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin L Ferguson, MD, Principal Investigator — University of Florida